CLINICAL TRIAL: NCT07241429
Title: Kinesiophobia, Balance Performance, Fear of Falling, and Related Factors in Stroke Patients
Brief Title: Kinesiophobia and Balance in Stroke Patients
Status: Recruiting | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Eser Kalaoglu, Principal Investigator, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Other Study IDs: IstPRMTRH-EK4
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Stroke
Keywords: Kinesiophobia; Postural Balance; Fear of Falling; Stroke
MeSH Terms: conditions — Stroke; Kinesiophobia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Inpatient Stroke Survivors: This observational group consists of 138 participants with a history of stroke (ischemic or hemorrhagic) who are receiving inpatient treatment at the Istanbul Physical Therapy and Rehabilitation Training and Research Hospital.
  Interventions: Other: Survey using a questionnaire.

INTERVENTIONS:
Other: Survey using a questionnaire. — All participants in this single cohort will undergo a one-time, cross-sectional assessment. This assessment includes the collection of clinical and demographic data and the administration of scales for kinesiophobia (Tampa Kinesiophobia Scale-17), balance performance (Berg Balance Scale), balance confidence (ABC-6), fear of falling (Falls Efficacy Scale), pain (VAS), and mood (HADS). No intervention is administered.

SUMMARY:
This is a cross-sectional clinical study planned to include 138 stroke patients receiving inpatient treatment at the Istanbul Physical Therapy and Rehabilitation Training and Research Hospital.Data on kinesiophobia (Tampa Kinesiophobia Scale-17) , balance performance (Berg Balance Scale) , balance confidence (Activities-specific Balance Confidence Scale-6) , fear of falling (Falls Efficacy Scale) , pain (VAS) , and mood (HADS) will be collected. Clinical and demographic data, including Brunnstrom stages and Barthel Index, will also be recorded. The relationships between these variables will be analyzed statistically.

DETAILED DESCRIPTION:
This is a cross-sectional clinical study planned to include 138 stroke patients receiving inpatient treatment at the Istanbul Physical Medicine and Rehabilitation Training and Research Hospital. Data on kinesiophobia (Tampa Kinesiophobia Scale-17) , balance performance (Berg Balance Scale) , balance confidence (Activities-specific Balance Confidence Scale-6) , fear of falling (Falls Efficacy Scale) , pain (VAS) , and mood (HADS) will be collected. Clinical and demographic data, including Brunnstrom stages and Barthel Index, will also be recorded. The relationships between these variables will be analyzed statistically

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation in the study
* Male and female patients aged 18-80
* History of ischemic or hemorrhagic stroke
* Functional Ambulation Scale level 3 or higher
* Standardized mini mental test ≥ 24
* Individuals who agree to participate in the study.

Exclusion Criteria:

* History of musculoskeletal surgery within the last year
* Trauma, fracture, dislocation, or tumor within the last year
* Vestibular system disorder
* Additional neurological disease that may affect balance (Parkinson's Disease, Multiple Sclerosis, vestibular system disorder)
* Other rheumatological or psychiatric diseases
* Chronic decompensated cardiac, renal, or hepatic failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The source population for this cross-sectional study is the adult patient population with a diagnosis of Stroke who are receiving inpatient physical medicine and rehabilitation services in a public training and research hospital setting in Turkey. Specifically, participants will be recruited from the İstanbul Physical Therapy and Rehabilitation Training and Research Hospital inpatient clinic. This setting provides access to a consecutive sample of individuals with varying degrees of functional deficits who are undergoing an organized rehabilitation program.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Estimated)
Dates: Start 2025-11-15 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of Kinesiophobia using the Tampa Kinesiophobia Scale-17 | at baseline assessment
  The Tampa Kinesiophobia Scale-17 (TKS-17) is a 17-item scale assessing fear of movement. It uses a 4-point Likert scale (1=Strongly disagree to 4=Strongly agree). Items 4, 8, 12, and 16 are reverse-scored. The total score ranges from 17 (minimum) to 68 (maximum). A higher score indicates a higher degree of kinesiophobia.

SECONDARY OUTCOMES:
Berg Balance Scale Score | at baseline assessment
  A 14-item scale assessing postural control. Each item is scored 0 (unable) to 4 (normal performance), with a maximum score of 56.
Falls Efficacy Scale Score | at baseline assessment
  A 10-item scale rating confidence in performing activities on a scale from 1 to 10. Total score ranges from 10 (minimum) to 100 (maximum). Higher scores indicate a higher level of fear of falling.
Hospital Anxiety and Depression Scale Score | at baseline assessment
  A 14-item scale with 7 items for anxiety and 7 for depression, each scored 0-3. Each subscale (Anxiety, Depression) has a maximum score of 21
Barthel Index Score | at baseline assessment
  Assessment of functional independence in activities of daily living.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Physical Therapy and Rehabilitation Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD), including all demographic, clinical, and primary/secondary outcome measures will be shared with qualified researchers. The sharing period will commence 6 months after article publication and conclude 1 year thereafter. Data access requests must be accompanied by a methodologically sound proposal and will be granted upon the corresponding author's approval and the execution of a Data Use Agreement (DUA) to strictly ensure confidentiality and adherence to ethical guidelines.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 6 months and ending 1 year following article publication.
Access Criteria: Qualified researchers who present a methodologically robust proposal aimed at fulfilling the objectives of the approved project.

REFERENCES:
- [Result] Pin TW, Winser SJ, Chan WLS, Chau B, Ng S, Wong T, Mak M, Pang M. Association between fear of falling and falls following acute and chronic stroke: a systematic review with meta-analysis. J Rehabil Med. 2024 Jan 16;56:jrm18650. doi: 10.2340/jrm.v56.18650. PMID 38226564
- [Result] Langhorne P, Bernhardt J, Kwakkel G. Stroke rehabilitation. Lancet. 2011 May 14;377(9778):1693-702. doi: 10.1016/S0140-6736(11)60325-5. PMID 21571152
- [Result] Batchelor FA, Mackintosh SF, Said CM, Hill KD. Falls after stroke. Int J Stroke. 2012 Aug;7(6):482-90. doi: 10.1111/j.1747-4949.2012.00796.x. Epub 2012 Apr 12. PMID 22494388